CLINICAL TRIAL: NCT03232489
Title: Open Label Study for the Evaluation of the Feasibility of Applying Advanced MRI Scanning in Pediatric Clinical Practice
Brief Title: Study for the Evaluation of the Feasibility of Applying Advanced MRI Scanning in Pediatric Clinical Practice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Principal Investigator, Sheldon Jordan, Neurologist, Neurological Associates of West Los Angeles
Other Study IDs: 20161363
Record Dates: First submitted 2017-06-12; First posted 2017-07-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to evaluate the feasibility in conducting advanced MRI sequences in a pediatric clinical setting. The study will be observational in nature, and will only evaluate the studies of pediatric patients who have already been prescribed an advanced MRI for clinical neurological purposes. The only difference for the subject in participating in this study is that the data and information about their scan can be used and disclosed for research purposes, i.e. understanding if the time of the scan, patient comfort, and quality of the data are feasible. Standard MRI's have been extremely beneficial in the diagnosis and assessment of disease, injury, and anomalies throughout the body. Adding advanced MRI sequences to the arsenal of current standard MRI sequences, as well as analyzing the clinical significance of the data, may improve the benefits of MRI in the future. Within this scope, the study will be looking at the following factors:

1. The total time of the scan, including:

   * Patient arrival time/lateness
   * Patient preparation time
   * Time scanner is being occupied
   * Patient compliance (is the patient continually stopping the study for breaks, fear, movement, etc.)
2. Patient dropout rate, including:

   * Change of mind
   * Cost of study is too much
   * Failure to finish the scan
3. Usability of data, including:

   * Movement artifact
   * Patient requiring re-scan for any reason

The scan will consist of two to five advanced MRI sequences that will average between 7-15 minutes each, in addition to a routine 5 minute standard MRI sequence. The variability in the number of advanced sequences depends on the prescription and patient history. All sequences are performed using a 1.5 Tesla Siemens MRI scanner at Westwood Open MRI, a 3 Tesla GE scanner at Tower Saint John's Imaging, or a 3 Tesla Siemens MRI scanner at Resolution Imaging. All scanners are FDA-approved.

DETAILED DESCRIPTION:
An MPRAGE is a high quality anatomical image of the brain. This is used as an anatomical overlay, so that all data collected from the advanced sequences below can be correlated with the correct brain areas in three-dimensional space.

1. Resting BOLD - BOLD stands for blood oxygen level dependent. This functional sequence allows for the viewing of the thinking brain at rest, and looks at brain areas that are functionally working together at the same time. The brain is in one of its most active states when it is at rest, and literature has shown that a few neurological illnesses such as OCD, depression, and pain have been associated with analyzing the data in this sequence.
2. Arterial Spin Labeling (ASL) - ASL tracks the blood flow in the brain visually and gives a statistical value of how much blood is in each region in cc's per 100 grams of brain per second.
3. Diffusion Tensor Imaging (DTI) - DTI tractography shows the different fiber tracts in the brain using a 3D model. Fiber tracts are the physical neural pathways that can show disruption or connection in communication between different areas of the brain. This is an effective technique when looking at traumatic brain injury.
4. Magnetic Resonance Spectroscopy (MRS) - MRS measures the ratios of select chemical compounds in the brain in relation to each other. This has shown to be effective in analyzing memory loss, dementia, and Alzheimer's type disorders.
5. Stimulated BOLD - The same sequence as the resting BOLD, except the brain is being scanned during the completion of a task, instead of rest. By specifying the task (visual, problem solving, language, etc.), the different areas of the brain working together to complete this task can be imaged. This is very effective for task-specific symptoms and deficits.

The methods and procedures in this study are all under the observational category. MRI's are FDA approved and are non-experimental devices. The goal of this research is to assess the feasibility of the scan itself, so everything done with respect to the scan is considered observational in nature. If the subject drops out of the study, anything described in this protocol will still be able available to the subject as standard medical care. The observational procedures will involve recording data for the advanced MRI scans, and no information will be shared for research if the subject does not sign the consent form.

ELIGIBILITY:
Inclusion Criteria:

In order for a subject to be considered for this study, the following criteria are required:

* The subject is between the ages of neonate-18 years old
* The subject clinically needs an advanced MRI
* The assent of the subject and the agreement of parent(s) or guardian(s) to the participation of their child or ward in research, in accordance with the regulations set forth in the Belmont Report

Exclusion Criteria:

In order for a subject to be considered for this study, he/she may NOT have any of the following items in which cannot be removed prior to the MRI exam. A subject that can remove any of the following prior to the MRI exam will still be considered for the study.

* Aneurism clips
* Cardiac pacemaker
* Implanted cardioinverter defibrillator
* Electronic implant or device
* Magnetically activated implant or device
* Neurostimulation system
* Spinal cord stimulator
* Internal electrodes or wires
* Bone growth/bone fusion stimulator
* Cochlear, otologic, or other ear implant
* Insulin or other infusion pump
* Implanted drug infusion device
* Any type of prosthesis (eye, penile, etc.)
* Heart valve prosthesis
* Eyelid spring or wire
* Artificial or prosthetic limb
* No Metallic stent, filter, or coil
* Shunt (spinal or intraventricular)
* Vascular access port and/or catheter
* Radiation seeds or implants
* Swan-Ganz or thermodilution catheter
* Medication patch (Nicotine, Nitroglycerine)
* Any metallic fragment or foreign body
* Wire mesh implant
* Tissue expander (e.g., breast)
* Surgical staples, clips, or metallic sutures
* Joint replacement (hip, knee, etc.)
* Bone/joint pin, screw, nail, wire, plate, etc.
* IUD, diaphragm, or pessary
* Dentures or partial plates
* Tattoo or permanent makeup
* Body piercing jewelry
* Hearing aid

As well as:

* Breathing problem or motion disorder
* Severe claustrophobia

Any subjects from the following categories/groups will NOT be included in the study:

* Prisoners
* Poor/uninsured
* Institutionalized
* Limited or non-readers
* Non-English speaking subjects
* Wards of the state
* Pregnant women
* Nursing home residents recruited in the nursing home
* Students of PI or study staff
* Students recruited in the educational setting (school, class, etc.)
* Employees directly supervised by the PI or sub-investigator
* Employees of research site or sponsor
* Military personnel recruited by military personnel
* Cognitively impaired
* Adult subjects that cannot consent for themselves

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects in this research study will be recruited by routine medical office exam.The ages for the subjects in this study will range from neonates to 18 years old.The gender distribution for this study will aim for a ratio of 50:50 male to female. There are no enrollment restrictions based upon race or ethnic origin. There are also no additional benefits, risks, advantages, or disadvantages based off of any race or ethnic origin.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-07; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects who successfully complete an fMRI scan | Through study completion, an average of 1 year
  In order to assess scan feasibility, we will keep track of the total number of patients who sign the consent form and are able to complete the fMRI scan.

SECONDARY OUTCOMES:
Subject appointment time vs. subject arrival time | Through study completion, an average of 1 year
  For each study subject, we will record the scheduled fMRI appointment time vs. the time that the subject arrives.
Time it takes subject to get from checked-in to start of scan (in minutes) | Through study completion, an average of 1 year
  For each study subject, we will record how long it takes to transition the subject from check-in to starting the fMRI scan.
How long was the scanner unoccupied (in minutes) | Through study completion, an average of 1 year
  We will record the length of time that the scanner is unoccupied in between scans.
Number and type of sequences performed | Through study completion, an average of 1 year
  For each study subject, we will record the number and type of sequences performed for the fMRI scan, e.g. MPRAGE, ASL, Resting BOLD, etc.
Time of scan (in minutes) | Through study completion, an average of 1 year
  For each study subject, we will record the total amount of time it takes to complete the fMRI scan.
How many times did the subject pause the scan (if any) and for how long (in minutes) | Through study completion, an average of 1 year
  For each study subject, we will record the number of times a subject pauses the fMRI scan and the duration of each pause.
Did the subject finish the scan | Through study completion, an average of 1 year
  For each study subject, we will record whether or not the subject was able to complete the fMRI scan.
Did the subject cancel the scan, and for what reason | Through study completion, an average of 1 year
  For each study subject, we will record whether the patient canceled the fMRI scan and for what reason.
Did the subject cause too much movement artifact | Through study completion, an average of 1 year
  For each study subject, we will record whether the post-processed fMRI data shows too much motion artifact, which could lead to the subject needing to be re-scanned.
Does the subject need to be re-scanned, and for what reason | Through study completion, an average of 1 year
  For each study subject, we will record whether or not the subject requires a re-scan and for what reason.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, MD, FAAN, Principal Investigator — Neurological Associates of West Los Angeles
Locations (1):
- Neurological Associates of West Los Angeles, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No